CLINICAL TRIAL: NCT04206085
Title: Comparison of the Viveve Treatment and Cryogen-Only Treatment Versus Sham Treatment for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viveve Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VI-19-01
Record Dates: First submitted 2019-12-10; First posted 2019-12-20 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2020-05

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Active treatment (Experimental): Radiofrequency and Cryogen
  Interventions: Device: Viveve - Active
- Cryogen-Only (Active Comparator): Crygen-Only
  Interventions: Device: Viveve - Cryogen-Alone
- Sham (Sham Comparator): Sham comparator
  Interventions: Device: Viveve - Sham

INTERVENTIONS:
Device: Viveve - Active — Radiofrequency and Cryogen-Cooling
  Arms: Active treatment
Device: Viveve - Cryogen-Alone — Cryogen-Cooling
  Arms: Cryogen-Only
Device: Viveve - Sham — Sham
  Arms: Sham

SUMMARY:
This is a prospective, randomized, single-blind, study comparing both the Viveve Treatment (RF plus cryogen) and cryogen alone treatment versus sham treatment in patients with mild to moderate stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal females, ≥ 18 years of age. Premenopausal is defined as a woman who has had menstrual cycles over the previous 12 months.
* Subjects with a BMI of ≤ 35 kg/m².
* 1-hr pad weight at Baseline with a 5 to 50 g net increase from the pre-test pad weight

Exclusion Criteria:

* Subjects who are currently breastfeeding or have discontinued breastfeeding fewer than 6 months prior to screening.
* Subjects who are pregnant or plan to become pregnant during the course of the study.
* Subjects who have undergone other stress urinary incontinence treatments, excluding behavioral modifications (e.g., Kegel exercises).
* Has any implantable electrical device [e.g., implantable pacemaker, automatic implantable cardioverter-defibrillator (AICD)].
* Subjects who have started or changed dose of local vaginal hormones <6 weeks before Screening.
* Subjects who have started pelvic floor physical therapy within the last 3 months.
* Undergone previous elective surgical or non-invasive procedure(s) in the vaginal canal (including the Viveve Treatment or any other genital radiofrequency treatment; injectable bulking agent, cosmetic, laser, surgical, and/or genital enhancement procedure, and previous dilation and cuterage within 12 months of the subject's Pre-Screening Visit).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 38 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Milestone Research, London, Ontario
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Devonshire Clinical Research, Woodstock, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment | Cryogen-Only | Sham
Started | 13 | 13 | 12
Completed | 13 | 12 | 11
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Cryogen-Only | Sham | Total
Number analyzed (Participants) | 13 | 13 | 12 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 12 | 38
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 12 in cryogen alone arm analyzed in full analysis set. 11 in sham arm analyzed in full analysis set.
  years
    number analyzed (Participants) | 13 | 12 | 11 | 36
    (all) | 42.6 (9.02) | 42.6 (7.38) | 43.3 (6.50) | 42.8 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 12 | 38
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 13 | 13 | 11 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 13 | 13 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: 1-hour Pad Weight Test
Description: Brief description of test:
  * Subject puts on one standardized, pre-weighed pad without voiding.
  * Subject drinks 500 mL of sodium-free liquid in < 15 min while sitting or resting.
    • 15 - 45 Minutes:
  * Subject walks for 30 minutes, including climbing one flight of stairs (up and down).
    • 45 - 60 Minutes:
  * Subject performs the following activities Standing up from sitting (10 times) Coughing vigorously (10 times) (Subject should be standing) Running on the spot (1 min) Bending to pick up an object from the floor (5 times) • The weight of the pad is measured to determine the amount of leakage.
Time Frame: Change in 1 hour Pad Weight Test Values at 5 Months from Baseline
Population: Full analysis set used.
Measure: Median (25% Confidence Interval); unit: Grams
Arm/Group | Active Treatment | Cryogen-Only | Sham
Number analyzed (Participants) | 13 | 12 | 11
Grams | -9.0 [-10.1 to -5.8] | -6.3 [-20.6 to -1.8] | -4.4 [-5.0 to 2.8]

ADVERSE EVENTS:
Time Frame: For each subject, adverse event collection occurred from treatment initiation at the randomization visit until the completion of the month 5 visit. The duration was 5 months.
Groups:
- Active Arm: 90 J/cm2 radiofrequency, 35 ms pulse cryogen cooling)
- Cryogen Arm: <1 J/cm2 radiofrequency, 35 ms pulse cryogen cooling
- Sham Arm: Completely inert tip
Arm/Group | Active Arm | Cryogen Arm | Sham Arm
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 8/13 | 2/13 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm (N=13) | Cryogen Arm (N=13) | Sham Arm (N=12)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Medical device site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic Discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT04206085/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT04206085/SAP_001.pdf